CLINICAL TRIAL: NCT05270434
Title: Optimal Timing of Endoscopic Intervention After Extracorporeal Shock-Wave Lithotripsy in the Treatment of Chronic Pancreatitis With Pancreatic Stones.
Brief Title: Optimal Timing of Endoscopic Intervention in the Treatment of Chronic Pancreatitis.
Acronym: TEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Optimal Timing of Endoscopic
Record Dates: First submitted 2022-01-10; First posted 2022-03-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pancreatitis, Chronic
Keywords: Extracorporeal Shock Wave Lithotripsy(ESWL); Chronic pancreatitis; Endoscopic Retrograde Cholangiopancreatography(ERCP); Pancreatic stones
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Cholangiopancreatography, Endoscopic Retrograde; Morphine; Buprenorphine; Meperidine; Dipyrone; Analgesics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic group <12h (Experimental): The patients received intravenous analgesia (flurbiprofen and remifentanil) before the ESWL (Compact Delta II; Dornier Med Tech, Wessling, Germany). After the last ESWL session, the patients are treated with following ERCP within 12h. ERCP was performed under conscious sedation with intramuscular administration of diazepam 2.5-5.0 mg and pethidine 25-50 mg. If necessary, endoscopic sphincterotomy was performed. A dilating bougie or balloon will be used to dilate the stenosis after sphincterotomy. Standard techniques (i.e., extraction basket, extraction balloon, or both) will be used for stone removal. A pancreatic duct stent for drainage and nasopancreatic catheters will be inserted for temporary drainage if necessary.
  Interventions: Procedure: time interval between ESWL and ERCP is 12h; Drug: morphine, buprenorphine, pethidine, tramaldol, metamizole and acetylsalicylacid (Analgesics)
- Endoscopic group ≥12 h (Active Comparator): The patients received intravenous analgesia (flurbiprofen and remifentanil) before the ESWL (Compact Delta II; Dornier Med Tech, Wessling, Germany). The time scale between the last ESWL session and following ERCP is greater than 12h. ERCP was performed under conscious sedation with intramuscular administration of diazepam 2.5-5.0 mg and pethidine 25-50 mg. If necessary, endoscopic sphincterotomy was performed. A dilating bougie or balloon will be used to dilate the stenosis after sphincterotomy. Standard techniques (i.e., extraction basket, extraction balloon, or both) will be used for stone removal. A pancreatic duct stent for drainage and nasopancreatic catheters will be inserted for temporary drainage if necessary.
  Interventions: Procedure: time interval between ESWL and ERCP is greater than 12h; Drug: morphine, buprenorphine, pethidine, tramaldol, metamizole and acetylsalicylacid (Analgesics)

INTERVENTIONS:
Procedure: time interval between ESWL and ERCP is 12h — The patients received intravenous analgesia before the ESWL. After the last ESWL session, the patients are treated with following ERCP within 12h.
  Other Names: ESWL; ERCP
  Arms: Endoscopic group <12h
Procedure: time interval between ESWL and ERCP is greater than 12h — The patients received intravenous analgesia before the ESWL. After the last ESWL session, the patients are treated with following ERCP ≥12 h.
  Other Names: ESWL; ERCP
  Arms: Endoscopic group ≥12 h
Drug: morphine, buprenorphine, pethidine, tramaldol, metamizole and acetylsalicylacid (Analgesics) — Analgesics administrated include morphine, buprenorphine, pethidine, tramaldol, metamizole and acetylsalicylacid. They will only be administrated as needed.

SUMMARY:
This study aims to determine the optimal timing of endoscopic intervention after extracorporeal shock wave lithotripsy(ESWL) of chronic pancreatitis with pancreatic stones.

DETAILED DESCRIPTION:
Chronic pancreatitis（CP）is a chronic progressive fibro-inflammatory disease of the pancreas induced by a wide range of factors including genetic and environmental elements, with recurrent abdominal pain and pancreatic secretion insufficiency as its major clinical signs. Chronic pancreatitis is not only a tough disease of the gastrointestinal system but also a worldwide medical problem. At present, the MESS (medicine-extracorporeal shock wave lithotripsy-endoscopic retrograde cholangiopancreatography-surgery）formed by changhai hospital in CP diagnosis and treatment is gradually becoming mature, and the clinical effect of this system is obvious. However, there are still some difficulties and knowledge gaps in the clinical treatment of CP. Currently, it is recommended by both domestic and foreign guidelines that ERCP combined with ESWL as the first-line treatment pattern for patients with chronic pancreatitis associate pain. It has previously been observed that ERCP performed less than 2 days after ESWL may be more likely to fail, possibly owing to ESWL-induced edema. However, there is no high-quality research to demonstrate how to choose the most optimal timing of ERCP after ESWL for patients with indications for endoscopic treatment. This prospective, randomized controlled research has therefore aimed to determine the most optimal timing of ERCP after ESWL. Patients with painful chronic pancreatitis and pancreatic stones larger than 5 mm in diameter will be randomly and equally assigned to two groups, which are divided according to the time interval between ESWL and ERCP, including the same day (< 12 hours) subgroup and the next day ( ≥12 hours) subgroup. The cannulation success rate and stone clearance rate of the pancreatic duct will be assessed in each group to explore the most appropriate timing of ERCP, and then provide an important reference basis for the clinical treatment of chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. symptomatic adult patients diagnosed with chronic pancreatitis and main pancreatic duct positive stones（>5mm in diameter）
2. no ERCP and ESWL history before the admission
3. provides informed consent

Exclusion Criteria:

1. suspected to have malignant tumors;
2. history of pancreatic surgery or gastrojejunostomy (Billroth II);
3. with end-stage disease;
4. with contraindications to ESWL or ERCP, such as pregnancy, abdominal aortic aneurysm, etc.
5. acute pancreatitis within 3 days
6. pancreatic ascites

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-10-18 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Successful MPD Cannulation Rates | during ERCP procedure
  technical success rate of pancreatic cannulation

SECONDARY OUTCOMES:
Successful clearance of MPD stones | during ERCP procedure
  Ductal clearance has been defined as complete, partial, or unsuccessful if the proportion of stones cleared was > 90 %, 50 %-90 %, or < 50 %, respectively.
post-ERCP complications | 30 days
  Major post-ERCP complications includes post-ERCP pancreatitis, bleeding, infection, and perforation, which are classified as mild, moderate, or severe, depending mainly on the length of hospitalization and the need for invasive treatment.
severity of post-ERCP complications | 30 days
  severity are classified as mild, moderate, or severe, depending mainly on the length of hospitalization and the need for invasive treatment.

OTHER OUTCOMES:
Treatment-related costs in RMB from initial enrollment to the end of the study | through endotherapy completion, an average of 14days
  The total costs in RMB of each hospitalization
The hospitalization time | through endotherapy completion, an average of 14days
  Length of hospitalization due to ESWL /ERCP and complications

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo JY, Qian YY, Sun H, Chen H, Zou WB, Hu LH, Li ZS, Xin L, Liao Z. Optimal Timing of Endoscopic Intervention After Extracorporeal Shock-Wave Lithotripsy in the Treatment of Chronic Calcified Pancreatitis. Pancreas. 2021 Apr 1;50(4):633-638. doi: 10.1097/MPA.0000000000001810. PMID 33939679